CLINICAL TRIAL: NCT06647784
Title: Effect of Lateralization Before and During Prone Position on Pulmonary Aeration During ARDS
Brief Title: Lateral Positioning and Prone Positioning in ARDS Patients
Acronym: LAT&PRONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Bastia (Other)
Collaborators: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LATPRON-24-01; ID-RCB 2024-A01321-46 (Other: ansm)
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: ARDS
Keywords: ARDS; Pulmonary aeration; Supine; prone position; lateralization
MeSH Terms: conditions — Deception | interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: Lateralization using a commercialy available bed (Multicare X LINET)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lateral and alterning positioning (Experimental): Baseline assessment in SP followed by repeated 30-minute lateral decubitus sessions on each side (with a 30° inclination) with a right/left alternation (total duration, 1 hour). During this period, the upper part of the bed will be inclined by 30°. The patients will then be positioned in prone position for a period of 6 hours after which, the same alternating lateral decubitus pattern (repeated 30-minute lateral decubitus sessions on each side with a right/left alternation ) will be applied for 12 hours while the patient is still in prone position. After turning back to the supine position, a 1-hour observation period will be respected before the last measurements are taken. The total duration of the intervention will thus be 20 hours.
  Interventions: Other: pulmonary aeration in supine and ventral decubitus

INTERVENTIONS:
Other: pulmonary aeration in supine and ventral decubitus — The addition of repeated periods of 30 minutes of lateralization of 30° amplitude in dorsal decubitus and in ventral decubitus in patients with moderate to severe ARDS. Included patients will benefit from sessions of lateral decubitus for 30 minutes on each side (with an inclination of 30°) with alternation right/left (total one hour). During this period, the upper part of the bed will be inclined by 30°. Patients will then be positioned in strict prone position for a period of 6 hours after which, the same pattern of alternating lateral decubitus will be applied for 12 hours while the patient is still in the prone position. After reversal in supine position, an observation period of 1 hour will be respected before carrying out the last measurements. The total duration of the intervention will be 20 hours.

SUMMARY:
Lateral (30°) and alternating positioning (change of side every 30 minutes) carried out on specific beds, could be an alternative or complement to prone positioning (PP) in ARDS patients. The combination of lateralization in prone position has not been studied. The dynamic created by lateralization could allow better overall ventilation during PP, thus making it possible to further improve oxygenation. The main objective of this prospective, bicentric, open, single group study with repeated measures will be to demonstrate that the addition of repeated 30-minute periods of 30° lateralization improves pulmonary aeration in the supine and prone positions in patients with moderate to severe ARDS.

DETAILED DESCRIPTION:
Primary objective: assessment of the distribution of tidal volume after lateralization and according to the position (supine position SP, prone position, PP) by measuring global and regional changes (4 regions of interest from the retrosternal region to the prevertebral region) of pulmonary aeration assessed by electrical impedance tomography (EIT). The primary endpoint will be the change in pulmonary aeration after lateralization in SP (T2) and in PP (T5) estimated by the change in end-expiratory lung impedance (EELI) = [ΔEELI x (VT/ΔZ)] where VT is the tidal volume and ΔZ is the impedance change.

Main secondary objective: assessment of perfusion and gas exchange after each period of lateralization compared to the baseline period in supine position (baseline SP) and in ventral position (baseline PP) (endpoints: PaO2/FiO2 and PaCO2)

Other secondary objectives:

* Evaluation of the percentage of patients who, at the end of the period of lateralization in supine position (T2), have a PaO2/FiO2 ratio > 150
* Comparisons baseline SP with baseline PP, PP 6 hours, PP and lateral positioning (LP) 12 hours and return to supine position since 1 hour (End) for pulmonary aeration, gas exchange and ventilatory parameters (endpoints: PaO2/FiO2 and PaCO2, (EELI) = [ΔEELI x (VT/ΔZ)], plateau pressure, driving pressure).
* Baseline PP comparisons with PP 6 hours, PP and lateral positioning (LP) 12 hours and return to supine position since 1 hour (End) for pulmonary aeration, gas exchange and ventilatory parameters (endpoints: PaO2/FiO2 and PaCO2, (EELI) = [ΔEELI x (VT/ΔZ)], plateau pressure, driving pressure)
* LP comparisons in SP for 6 hours with LP in PP for 12 hours for pulmonary aeration, gas exchange and ventilatory parameters (endpoints: PaO2/FiO2 and PaCO2, (EELI) = [ΔEELI x (VT/ΔZ)], plateau pressure, driving pressure)
* LP comparisons in PP for 12 hours with return to supine position since 1 hour (End) for pulmonary aeration, gas exchange and ventilatory parameters (endpoints: PaO2/FiO2 and PaCO2, (EELI) = [ΔEELI x (VT/ΔZ)], plateau pressure, driving pressure) : PaO2/FiO2 and PaCO2, (EELI) = [ΔEELI x (VT/ΔZ)], plateau pressure, driving pressure)
* Evaluate the adverse effects related to the use of lateral positioning.

ELIGIBILITY:
Inclusion criteria:

* Age of at least 18 years
* ARDS evolving for less than 5 days with a PaO2/FiO2 ratio (P/F ratio) < 150 after optimization of PEEP (P/V curve, R/I ratio), curarization and without prior use of the PP since orotracheal intubation.
* Obtained written consent of the patient, one of his relatives or the previously designated trusted person. As soon as possible, the patient will be informed and his written consent will be obtained
* Beneficiary of health insurance coverage
* Possibility of participating in any other studies whose evaluation criteria do not interfere with those of the study

Non-inclusion criteria:

Patients with at least one of the following criteria will not be eligible:

* Refusal to participate
* Pregnant, parturient or breastfeeding women
* Intracranial pressure > 30 mm Hg or cerebral perfusion pressure < 60 mmHg
* Severe chronic respiratory disease with oxygen therapy or mechanical ventilation at home (except CPAP/BIPAP for obstructive sleep apnea)
* Chronic interstitial lung diseases
* Patients on ECMO
* Weight > 100 kg
* Severe liver disease Child-Pugh score 12-15
* Pneumothorax
* SAPS II score > 75 at inclusion
* Unstable spinal fracture
* Contraindications to EIT (pacemaker, implantable defibrillator, skin lesions between the 4th and 5th ribs).
* Withdrawal (except for ECMO) or witholding treatment decision
* Any other reason which, according to the investigator, could interfere with the evaluation of the study objectives
* Person under legal protection measure (guardianship, curatorship, etc.)
* Person deprived of liberty by a judiciary or administrative decision

Exclusion criteria:

- Patients who will be unable to complete the 25-hour intervention due to worsening requiring ECMO, death or organizational problems will be excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
modification of pulmonary aeration | Up to 25 hours.
  Evaluation of the distribution of tidal volume after lateralization and according to the position (supine: SP, prone: PP) by measuring global changes and regional (4 regions of interest from the retro-sternal region to the pre-vertebral region) of ventilation lung assessed by electrical impedance tomography (EIT).The primary endpoint will be the change in pulmonary aeration after lateralization in SP (T2) and in PP (T5) estimated by the variation in end-expiration pulmonary impedance (EELI) = [ΔEELI x (VT/ΔZ)] where VT is the tidal volume and ΔZ the impedance variation.

SECONDARY OUTCOMES:
Assessment of gas exchange | Up to 25 hours
  Assessment of gas exchange (by blood gas analyses) after each each lateralization period compared with the baseline period in dorsal position (SP) and prone position (baseline PP) (endpoints: PaO2/FiO2 and PaCO2)
Assessment of lung perfusion | Up to 25 hours
  Assessment of lung perfusion by EIT (administration of 10 ml 7.5% hypertonic saline during an expiratory pause)

OTHER OUTCOMES:
Estimated PaO2/FiO2 ratio > 150 | Up to 25 hours
  Evaluation of the percentage of patients with a PaO2/FiO2 ratio > 150 at the end of the supine lateralization period
Measurement of lung aeration | Up to 25 hours
  Comparisons of : baseline SP with baseline PP, 6-hours PP, PP and lateral positioning (LP) 12h and return to supine for 1h (End), baseline PP with PP 6 hours, PP and lateral positioning (LP) 12h, LP in SP for 6h with LP in PP for 12h and LP comparisons in PP for 12h with return to supine for 1h (End) for pulmonary aeration, (endpoints: PaO2/FiO2 and PaCO2, (EELI) = [ΔEELI x (VT/ΔZ)], plateau pressure, driving pressure).
Gas exchange assessment | Up to 25 hours
  Comparisons of baseline SP with baseline PP, 6-hours PP, PP and lateral positioning (LP) 12h and return to supine for 1h (End), baseline PP with PP 6 hours, PP and lateral positioning (LP) 12h, LP in SP for 6h with LP in PP for 12h and LP comparisons in PP for 12h with return to supine for 1h (End) for gas exchanges (endpoints: PaO2/FiO2 and PaCO2).
Measurement of ventilatory parameters | Up to 25 hours
  Comparisons of baseline SP with baseline PP, 6-hours PP, PP and lateral positioning (LP) 12h and return to supine for 1h (End), baseline PP with PP 6 hours, PP and lateral positioning (LP) 12h, LP in SP for 6h with LP in PP for 12h and LP comparisons in PP for 12h with return to supine for 1h (End) for ventilatory parameters (plateau pressure, driving pressure, compliance, elastance).
Adverse effects | Up to 25 hours
  Evaluate adverse effects associated with the use of lateral positioning.

CONTACTS AND LOCATIONS:
Overall Officials: laurent papazian, MD,PHD, Study Director — Bastia General Hospital
Locations (2):
- France (2):
  - Bastia General Hospital, Bastia, France
  - North Hospital Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: When the study will be completed
Access Criteria: To be determined when the study will be completed